CLINICAL TRIAL: NCT07078383
Title: Evaluation of the Rapidlink Device for Use in the Repair or Replacement of the Supra-Aortic Vessels During an Open Surgical Procedure of the Thoracic Aorta
Brief Title: A Study to Evaluate the Safety and Effectiveness of the Rapidlink Device When Used in Patients Undergoing an Open Surgical Procedure to Repair the Aorta
Acronym: RAPID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPID-001
Record Dates: First submitted 2025-06-19; First posted 2025-07-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Aortic Aneurysm; Aortic Aneurysm and Dissection; Aortic Diseases; Aneurysm of Aorta, Thoracic; Aneurysmal Disease; Aorta, Thoracic Pathologies
Keywords: Vascular Prosthesis; Replacement or bypass of disease vessels; aneurysmal disease; Aortic branch vessels; Open aortic arch repair; aneurysm; dissection; Supra-aortic Vessels; Frozen Elephant Trunk; Left Subclavian Artery
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Aortic Diseases; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Rapidlink Device (Experimental)
  Interventions: Device: Rapidlink

INTERVENTIONS:
Device: Rapidlink — The Rapidlink implant is comprised of a Gelweave graft section (gelatin-sealed woven polyester) attached to a stented section (which utilizes nitinol ring stents), with a 'cuff'' feature joined to the stented section of the implant. The implant is supplied pre-loaded in a single use delivery system which compacts the stented section within a polytetrafluoroethylene (PTFE) sheath at the front of the system.

SUMMARY:
The Goal of this Clinical Study is to evaluate the safety and effectiveness of the Rapidlink device in the repair or replacement of the supra-aortic vessels during open surgical repair of aortic disease affecting the thoracic aorta.

This study will collect information on patients who are already having surgery to repair their aorta and who will have Rapidlink device implanted into one or more of the aortic arch vessels.

The first 32 subjects enrolled will undergo left subclavian artery repair or replacement, only, with the Rapidlink device. After the 32nd subject, enrollment will proceed to include subjects undergoing any supra-aortic vessel (i.e., left subclavian artery, left common carotid artery, and/or innominate artery) repair or replacement with the Rapidlink device in a planned surgery.

After the 32nd subject is enrolled in the main group, up to 30 subjects will undergo supra-aortic vessel (i.e., left subclavian artery, left common carotid artery, and/or innominate artery) repair or replacement with the Rapidlink device in an emergency setting.

Data will be collected before, during and after surgery including recovery at discharge, 30 days, 6 months, 1 and 2 years after the surgery.

DETAILED DESCRIPTION:
Treatment options for pathologies involving the aortic arch include medical management, open surgical repair with vascular grafts (e.g., Gelweave), and frozen elephant trunk procedures (e.g., Thoraflex Hybrid).

During conventional replacement of the aortic arch, branches from the main graft are anastomosed onto the transected main arch vessels. In some circumstances this can be difficult for the surgeon, particularly in the case of the left subclavian artery which can be deep routed and difficult to access due to patient anatomy. It can also be displaced by aneurysmal disease or be fragile and friable secondary to atherosclerotic change.

An unmet need exists regarding the ability to access the supra-aortic vessels (e.g., left subclavian artery) in a timely manner during open surgical repair and to expedite the anastomosis to the arch while reducing the need to perform additional concomitant procedures (e.g., transposition or bypass of the left subclavian artery).

The Rapidlink device is designed to simplify this process by enabling the surgeon to place a stented graft within the supra-aortic vessels and secure it, with minimal sutures and manipulation, in a timely manner during open surgical repair.

This study will evaluate patients necessitating repair or replacement of the supra-aortic vessels (i.e., left subclavian artery, left common carotid artery, and/or innominate artery) during open surgical repair of aortic disease affecting the thoracic aorta in an elective (Primary Arm) or emergent (Emergent Arm) setting

Up to 120 subjects will be recruited in the primary arm (elective setting).The first 32 subjects will undergo left subclavian artery repair or replacement with the Rapidlink device. After the 32nd subject with only the left subclavian artery repair or replacement with the Rapidlink device has been enrolled, enrollment will proceed to include subjects undergoing any supra-aortic vessel (i.e., left subclavian artery, left common carotid artery, and/or innominate artery) repair or replacement with the Rapidlink device in an elective setting.

For the Emergent Arm, up to 30 subjects will undergo supra-aortic vessel (i.e., left subclavian artery, left common carotid artery, and/or innominate artery) repair or replacement with the Rapidlink device in an emergent setting. Enrollment into the Emergent Arm will begin after the 32ndsubject from the Primary Arm has been enrolled. Investigators are not allowed to enroll into the Emergent Arm until one elective case has been performed.

It is anticipated that up to 150 patients will be recruited over a 12 month period (approximately). Patients will be evaluated at the following timepoints: Pre-procedure, Implant, Discharge/30 days, 3 months, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years or over on date of consent
* Written informed consent (from patient or a legally authorized representative) to participate in study, documenting willingness and ability to comply with all study procedures and study visits (unless an exemption for emergency cases has been IRB / EC approved)
* Patient's need for open surgical repair of the thoracic aorta using a Gelweave graft or a Thoraflex Hybrid device (AnteFlo or Plexus) in line with the applicable IFU
* Anticipated need to use Rapidlink for the repair or replacement of the LSA, LCCA and/or IA during the open surgical repair
* Patient has an 8-15 mm inner diameter (target SAV)
* The diameters of the patient's target supra-aortic vessel(s), fall within the ranges specified in the IFU

Exclusion Criteria:

* Patient does not have a clear landing zone equal to the implantable stent length which is free from stenosis, calcification or thrombus.
* Patient does not have a sealing zone free from tortuosity.
* Patient has significant angulation (>79° with an internal radius of less than 6mm) for the full implantable stent length
* Patient cannot receive anticoagulation / antiplatelet therapy during or after the index procedure as per the protocol
* Patient has uncontrolled hypercoagulation
* Patient has a condition which may compromise or prevent the necessary imaging requirements
* Patient has anatomic variants which would compromise circulation to the first branch off the target artery after placement of the Rapidlink device (unless planned and/or otherwise revascularized)
* Patient is unfit for open surgical repair involving circulatory arrest per the study investigator
* Patient has known sensitivity to polyester, nitinol, tantalum, or materials of bovine origin
* Patient has a ruptured aorta
* Patient has active endocarditis or an active infective disorder of the aorta
* Patient has an active systemic infection that, in the opinion of the investigator, would compromise the outcome of the surgical procedure
* Patient is enrolled in another active study and has received an investigational product (device, pharmaceutical or biologic) within 6 months prior to the date of the implant or has not reached the primary endpoint of the study
* Patient is female and is pregnant or planning to become pregnant during the course of the study. Females of childbearing potential must use acceptable methods of contraception during the course of the study.
* Patient has an uncorrectable bleeding anomaly
* Patient has renal failure (defined as dialysis dependent or serum creatinine ≥2.5mg/dL)
* Patient has known sensitivity to radiopaque contrast agents that cannot be adequately pre-treated
* Patient has a co-morbidity causing expected survival to be less than 1 year
* Patient has any other medical, social or psychological problems that in the opinion of the investigator preclude them from receiving this treatment and the procedures and evaluations pre and post procedure
* Patient has a known chronic aortic dissection involving the intended landing zone of the target supra-aortic vessel(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
The absence of a major adverse event (MAE) at 6-month post procedure. | 6 months post procedure
  The primary endpoint is the absence of a major adverse event (MAE) at 6-month post procedure. MAE are defined as follows are will be assessed as composite and individually:
  Permanent disabling stroke Permanent paraplegia/paraparesis Device-related (Rapidlink) reinterventions All-cause mortality
  * Device-related mortality (arch graft and/or branch graft)
  * Procedure-related mortality
  * Not device or procedure related

SECONDARY OUTCOMES:
Technical Success of the Rapidlink portion of the procedure | 30 days post-procedure
  Technical Success: of the Rapidlink portion of the procedure is a composite endpoint evaluated at 30 days by the implanting physician and is defined as follows:
  * Successful access to the arterial system
  * Successful delivery and deployment of the Rapidlink device in the planned location without unplanned vessel coverage
  * Absence of Rapidlink-related Type I or Type III endoleaks (or resolution by 30 days) as determined by imaging confirmation
  * Patency of the Rapidlink device (defined as less than 50% stenosis or without the need for re-intervention due to stenosis),
  * Absence of device deformations requiring unplanned placement of an additional device
  * Successful withdrawal of the Rapidlink delivery system (without unanticipated corrective action related to the withdrawal)
Clinical Success (Total Arch Repair) | At discharge/30 days, 6-Months, 12 Months and 24 Months post-procedure
  Clinical Success (Total Arch Repair) is defined as:
  * Absence of lesion-related mortality
  * Absence of persistent Type I or Type III endoleak*
  * Absence of device infection
  * Absence of aortic thrombosis
  * Absence of new dissection
  * Absence of loss of patency (any unanticipated loss of patency of supra-aortic vessels)**
  * Absence of secondary intervention or conversion to open surgery completed to address a loss of device integrity
  * Absence of permanent paraplegia/paraparesis, permanent stroke, or laryngeal nerve paralysis that resulted from the initial operation or a secondary intervention to correct the treated supra-aortic vessels connections
  Clinical Success will be assessed as a composite and all individual elements
Rate of Aortic or supra-aortic vessel rupture | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Rate of Aortic or supra-aortic vessel rupture
Rate of Stroke of any type, including transient ischemic attacks | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Rate of Stroke of any type, including transient ischemic attacks
Rate of Pseudoaneurysm in the treated segment | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Rate of Pseudoaneurysm in the treated segment of the aorta
Device-related serious adverse events | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Rate of Device-related serious adverse events
Rate of endoleaks | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Rate of core laboratory imaging confirmed endoleak of any type
Rate of migration of the Rapidlink Device | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Migration defined as: Movement (caudal and/or cranial) of device of >10 mm as compared to first post-procedural imaging (e.g., discharge/30-day).
Rate of Loss of Device (Rapidlink) integrity | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Fracture of stent and or disruption of fabric or suture material as confirmed by imaging.
Patency related observations (e.g., asymptomatic loss of patency, stenosis) of the Rapidlink device | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Rate of patency related observations by type, confirmed by imaging
Rate of Lesion or device-related secondary interventions | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Rate of lesion or device-related secondary interventions
Clinical utility measures | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Duration of procedure and Implantation of Device (Hours)
Clinical utility measures | At discharge/30 days, 6-months, 12 months and 24 months post-procedure
  Volume of Bloodloss and Volume of transfusion or replacement blood products
Clinical Utility Measures | At discharge/30days, 6 months, 12 months and 24 months post-procedure
  Length of Duration of hospital stay (days)
Clinical Utility Measures | At discharge/30days, 6 months, 12 months and 24 months post-procedure
  Duration in Intensive Care Unit (days)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (16):
  - Keck Medicine of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Acension Seton Medical Center, Austin, Texas
  - Baylor Scott & White The Heart Hospital - Plano, Plano, Texas
  - Froedhert Hospital, Milwaukee, Wisconsin
- University Hospital Vienna, Vienna, Austria
- Germany (3):
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Robert Bosch Hospital, Stuttgart
- Radboud University Medical Center, Nijmegen, Radboud, Netherlands
- University Hospital of Bern, Bern, Switzerland
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided